CLINICAL TRIAL: NCT06024044
Title: The Effect of Mobilization Training Given to Women Before the Hysterectomy Operation on Post-Operational Bottom Functions and Pain: A Randomized Controlled Study
Brief Title: Effect of Mobilization Training Given to Hysterectomy Operation on Bottom Functions and Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, Burcu KUCUKKAYA, Assist. Prof, Bartın Unıversity
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2022/P428
Record Dates: First submitted 2023-08-29; First posted 2023-09-05 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Mobilization; Training Group
Keywords: Hysterectomy; Women; Post-Operational; Bottom Functions; Pain; Mobilization Training
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): The women patients in the control group who underwent hysterectomy were informed that mobilization training would be performed after a postoperative 2-day waiting period. Meanwhile, no intervention was made except for any routine nursing care.
- Mobilization Training (Experimental): A face-to-face "Patient Information Form" was applied to the training group in the first interview before the hysterectomy operation. The participants in the training group were given hysterectomy postoperative mobilization training by the researcher (B.K) using presentation and verbal information technique. A "Post-Operative Follow-up Chart" was given to the participants to fill in the 1st and 2nd postoperative days. The training group participants were followed up by the researcher on the 0th and 1st days after the operation in line with the mobilization training they received. The "Post-Operative Follow-up Chart" questioning the patients' mobilization times, distances, bowel functions and pain scores was filled in by the researcher in detail by face-to-face interview method. Mobilization time (minutes) and distance (meters) were evaluated by the patients and their relatives, and recorded on the chart, using the stopwatch and pedometer on the personal mobile phones of the patients.
  Interventions: Behavioral: Mobilization Training

INTERVENTIONS:
Behavioral: Mobilization Training — The participants in the training group were given hysterectomy postoperative mobilization training by the researcher (B.K) using presentation and verbal information technique. A "Post-Operative Follow-up Chart" was given to the participants to fill in the 1st and 2nd postoperative days. The training group participants were followed up by the researcher on the 0th and 1st days after the operation in line with the mobilization training they received. The "Post-Operative Follow-up Chart" questioning the patients' mobilization times, distances, bowel functions and pain scores was filled in by the researcher in detail by face-to-face interview method. Mobilization time (minutes) and distance (meters) were evaluated by the patients and their relatives, and recorded on the chart, using the stopwatch and pedometer on the personal mobile phones of the patients.
  Arms: Mobilization Training

SUMMARY:
Objectives: Research on the effect of mobilization training given to women before the hysterectomy operation on post-operational bottom functions and pain is a new and promising feld of research. However, high-level evidence on whether mobilization and mobilization training has an effect on bowel function and pain is insufficient. The present study addresses this research question.

Design: A two-arm randomized controlled trial was conducted in 82 women patients.

DETAILED DESCRIPTION:
This two-arm randomized controlled trial (RCT) was conducted in the women patients undergoing hysterectomy located in Edirne, between May 2022 and June 2023. During the intake, the women patients undergoing hysterectomy were informed about the goals and setup of the study and intervention, and assessed for eligibility by a brief standardized interview. The women patients undergoing hysterectomy who fulfilled our criteria received an information letter and informed consent form, as well as the baseline questionnaire. Those women patients undergoing hysterectomy that provided written informed consent for participation were included in the study. Assessments in both groups were performed before randomization (i.e., baseline) and directly after the intervention period.

Randomization: The women patients undergoing hysterectomy were randomly assigned to an education or control groups. A research assistant not actively involved in the design and data analysis of the study created a random distribution sequence and assigned participants to one of the two conditions (1:1 ratio).

Intervention:

Mobilization Training: A face-to-face "Patient Information Form" was applied to the training group in the first interview before the hysterectomy operation. The participants in the training group were given hysterectomy postoperative mobilization training by the researcher (B.K) using presentation and verbal information technique. A "Post-Operative Follow-up Chart" was given to the participants to fill in the 1st and 2nd postoperative days. The training group participants were followed up by the researcher on the 0th and 1st days after the operation in line with the mobilization training they received. The "Post-Operative Follow-up Chart" questioning the patients' mobilization times, distances, bowel functions and pain scores was filled in by the researcher in detail by face-to-face interview method. Mobilization time (minutes) and distance (meters) were evaluated by the patients and their relatives, and recorded on the chart, using the stopwatch and pedometer on the personal mobile phones of the patients.

Control Group: The women patients in the control group who underwent hysterectomy were informed that mobilization training would be performed after a postoperative 2-day waiting period. Meanwhile, no intervention was made except for any routine nursing care.

Measures: "Patient Information Form" and "Post-Operative Follow-up Chart" were used in the study. Patient Information Form: It was created by the researchers by scanning the literature and consists of a total of 18 questions, including 6 questions about the personal characteristics of the participants, 3 questions about the obstetric and surgical characteristics, and 9 questions about the postoperative results. Postoperative Follow-up Chart: It was created by the researchers by scanning the literature and consists of a 24-hour chart including the 0 and 1 postoperative day mobilization time, mobilization distance, pain score, gas and stool output time of the participants.

Sample size calculation for the primary research question was performed based on a pilot study. Tharwat et al. (2021), within the scope of the findings of their study named "Impact of Sugarless Chewing gum Versus Peppermint on First Bowel Movement after Cesarean Section: Randomized Controlled Trial", sample calculation was made by predicting the effect size of 0.6307060, 95% confidence level, and 80% power. Power analysis of the study was performed with G*POWER 3.1.9.7 (Power analysis statistical software) program (Faul et al., 2021). A total of 82 women with hysterectomy (Training group: 41 women, Control group: 41 women) constituted the sample.

ELIGIBILITY:
Inclusion Criteria:

* Having hysterectomy surgery,
* At least primary school graduate,
* With good mental functions,
* Not experiencing serious depression, anxiety and stress,
* No serious postoperative complications,
* No chronic pain,
* No sensory problems (vision loss, auditory loss, etc.),
* Women who volunteered to participate in the study.

Exclusion Criteria:

* Diagnosed with depression, anxiety and stress disorder,
* Diagnosed with chronic pain,
* Women who did not volunteer to participate in the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The women patients undergoing hysterectomy
Enrollment: 82 (Actual)
Dates: Start 2022-05-12 (Actual); Primary Completion 2022-05-14 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
Pain evaluated using the Visual Analog Scale | change from baseline implamentation patent and after 0 and 1 postoperative day of practice.
  The intensity of pain is measured using the VAS, a valid and reliable tool for measuring experimental and clinical pain. The VAS is scored on a horizontal line of 10 cm (0=no pain and 10=worst possible pain).

SECONDARY OUTCOMES:
Bottom functions evaluated using the Postoperative Follow-up Chart | change from baseline implamentation patent and after 0 and 1 postoperative day of practice.
  It was created by the researchers by scanning the literature, and consists of a 24-hour chart including the 0 and 1 postoperative day mobilization time, mobilization distance, pain score, gas and stool output time of the participants.

CONTACTS AND LOCATIONS:
Overall Officials: Burcu Küçükkaya, Asst. Prof., Principal Investigator — Bartın University, Faculty of Health Sciences, Nursing Department, Division of Gynecology and Obstetrics Nursing, Bartın, Turkiye; Zeynep Kızılcık Özkan, Asst. Prof., Principal Investigator — Trakya University, Faculty of Health Sciences, Nursing Department, Division of Surgery Nursing, Edirne, Turkiye
Locations (1):
- Trakya University, Edirne, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided